CLINICAL TRIAL: NCT03918343
Title: Study of Lipopolysaccharide Metabolism for Identification of New Biomarkers Predictive of Graft-versus-host Disease After Allogeneic Stem Cell Transplantation
Brief Title: Lipopolysaccharide Metabolism and Identification of Potential Biomarkers Predictive of Graft-versus-host Disease After Allogeneic Stem Cell Transplantation
Acronym: MetAlloLip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2018/387
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Diseases; Stem Cell Transplantation
MeSH Terms: conditions — Hematologic Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Other)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — blood samples (4 times; 14ml per visit)

SUMMARY:
This study is designed to assess the hypothesis that the lipopolysaccharide (LPS) activity index can be quantified early after transplantation, as well as the the PhosphoLipid Transfer Protein (PLTP) activity and these both biological variables are independent variables for predicting the risk of severe Graft versus Host Disease (GVHD).

ELIGIBILITY:
Inclusion Criteria:

* Hematologic malignancy in complete remission
* Patients eligible for allogeneic hematopoietic cell transplantation from a related or unrelated donor and after myeloablative or non-myeloablative conditioning.
* Regular follow-up in the center

Exclusion Criteria:

* Treatment with a statin in progress
* Umbilical cord blood transplantation
* Hemoglobin level less than or equal to 8g / dl
* Known chronic inflammatory bowel disease or gastroenteritis at the time of inclusion.
* Chronic enteropathy with Clostridium Difficile

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2025-05-23 (Actual)

PRIMARY OUTCOMES:
Area under the ROC curve for PLTP in the occurrence of GVHD | 3 months
  Area under the ROC curve (AUCROC) for PLTP assessed at day 0 (day of transplantation) in the occurrence of GVHD (grade II-IV) at 3 months post-transplant.
Area under the ROC curve for LPS in the occurrence of GVHD | 3 months
  Area under the ROC curve (AUCROC) for LPS assessed at day 0 (day of transplantation) in the occurrence of GVHD (grade II-IV) at 3 months post-transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Daguindau, MD, Principal Investigator — CHU Besançon
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire de Besançon, Besançon
  - Centre Hospitalier Universitaire de Nancy, Nancy

IPD SHARING:
Plan to Share IPD: No